CLINICAL TRIAL: NCT06351384
Title: Early Detection and Risk Stratification of Colorectal Cancer Based on miRNA Platform: a Prospective, Pilot Study
Brief Title: Early Detection and Risk Stratification of Colorectal Cancer Based on miRNA Platform
Status: Not yet recruiting | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20230744
Record Dates: First submitted 2024-04-01; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Colorectal cancer arm
  Interventions: Device: miRNA detection test
- Healthy control arm
  Interventions: Device: miRNA detection test
- Intestinal polyp arm
  Interventions: Device: miRNA detection test

INTERVENTIONS:
Device: miRNA detection test — miRNA sequencing based on Next-Generation Sequencing (NGS) technology

SUMMARY:
This is a prospective, observational cohort study to establish the minimal residual disease (MRD) model for predicting relapse risk and identifying disease recurrence in patients with colorectal adenocarcinoma based on the miRNA platform.

Blood miRNA markers will be evaluated. The study will enroll approximately 600 participants, including participants with malignancies or benign diseases, and healthy participants.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for the colorectal cancer arm:

1.18-75 years old 2. Pathologically confirmed as colorectal adenocarcinoma 3. Medically able to receive radical surgery for colorectal cancer 4. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 to 1 5. Ability to provide a written informed consent

Inclusion Criteria for the healthy control arm:

1.18-75 years old 2. No clinically significant finding based on routine blood tests, urinalysis, CT, and ultrasound examinations 3. Ability to provide a written informed consent

Inclusion Criteria for the intestinal polyp arm:

1.18-75 years old 2. Pathologically confirmed as colorectal adenoma 3. Ability to provide a written informed consent

Exclusion Criteria:

1. History of other malignant tumors (excluding non-melanoma skin cancer).
2. Prior or related treatments previously (including colorectal cancer or advanced adenoma surgery, endoscopic treatment, chemotherapy, targeted therapy, immunotherapy, radiation, neoadjuvant therapy, etc.).
3. Patients with hereditary colorectal diseases (including Lynch syndrome, familial CRC type X (FCCX), familial adenomatous polyposis (FAP), MUTHY-associated polyposis (MAP), Peutz-Jeghers syndrome (PJS), juvenile polyposis syndrome (JPS), serrated polyposis syndrome (SPS), etc.).
4. Usage of anti-tumor drugs such as methotrexate, cyclophosphamide, mercaptopurine, and bendamustine for other diseases within 30 days before blood collection.
5. Prior blood transfusion (including blood components) within the past 2 weeks.
6. Prior organ transplantation, bone marrow transplantation, or stem cell transplantation.
7. Pregnancy women.
8. Acute inflammation or fever requiring drug escalation within 14 days prior to blood collection.
9. Inability to comply with study procedures such as blood collection and related examinations.
10. Deemed unsuitable for participation in the clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from medical centers and assigned into three arms, including participants with new diagnosis of colorectal adenocarcinoma, participants with intestinal polyp, and healthy control.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between post-surgery 1 month MRD status and recurrence-free survival (RFS) in colorectal patients | 24 months

IPD SHARING:
Plan to Share IPD: No